CLINICAL TRIAL: NCT01950494
Title: A One Month, Randomized, Two-center, Parallel-group, Double-blind,Placebo-controlled Study to Evaluate the Efficacy and Safety of FiteBac Hand Sanitizer TID vs Emollient Therapy in the Management of Hand Dermatitis in Adults
Brief Title: FiteBac Hand Sanitizer in the Management of Hand Dermatitis in Adults
Acronym: FiteBac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Donald Leung, MD, PhD, Principal Investigator, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FiteBacFINAL; Fite Bac Hand Sanitizer (Other: FiteBac Hand Sanitizer)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Hand Dermatitis
Keywords: hand dermatitis; health care workers; hand sanitizer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fiteBac Hand Sanitizer (Experimental): Blinded fitBac Hand sanitizer
  Interventions: Other: fiteBac Hand Sanitizer
- Blinded emollient therapy (Placebo Comparator): Blinded emollient therapy
  Interventions: Other: fiteBac Hand Sanitizer

INTERVENTIONS:
Other: fiteBac Hand Sanitizer — Skin gel created for health care workers that is currently on the market. This sanitizer has an additive layer to protect the skin that is also thought to helpo hand dermatitis.
  Other Names: Brand name: fiteBac Hand Sanitizer

SUMMARY:
Hand dermatitis, (a rash, or eczema, on the hands) is a common skin condition that affects approximately 10% of the population. It can be caused by a wide variety of things, such as allergens or irritants. For some, it can be painful and disfiguring. In moderate to severe cases, hand dermatitis can interfere greatly in the quality of life of the affected person, interfering with work and social functions. This can have a negative psychological effect as well.

FiteBac Skin Care Gel is a new over-the-counter hand sanitizer that has been used for hospital and dental hand infection control. This product contains a germicide, to prevent infection. It also contains a silicone polymer. This makes the hand gel more durable, causing it to remain on the skin longer. Despite this durability, the hand gel still allows the skin to naturally perspire (sweat).

As people in the health-care industry have used this new product with the goal of reducing hand infections, it has been noted that FiteBac Skin Care Gel also seems to have reduced hand dermatitis and improved personal skin condition. The purpose of this study is to scientifically measure skin improvement in a population of study subjects with hand dermatitis.

DETAILED DESCRIPTION:
1. Informed consent must be signed and understood by subject.
2. Symptoms and history consistent with hand dermatitis based on symptoms and clinical history (as described in refs 4-7).
3. Males or females, 18-70 years of age, in generally good health with no significant underlying systemic disease requiring ongoing medications.
4. Hand eczema severity index (HECSI) with a score of greater than 50 (see Table 1 and reference 5)
5. Physician global assessment (PGA) of moderate to severe (with PGA severity scores graded as in Table 1 of reference 8: severe, moderate, mild, almost clear, clear).

3.2.3. Exclusion criteria

1. Topical corticosteroid or calcineurin inhibitor treatment during the last 7 days, prior to enrollment, on the hands and forearms
2. Systemic treatment with corticosteroids or other immunosuppressives during the last 14 days.
3. Subjects currently receiving (or received during the previous 4 weeks) other investigational drugs, treatments or devices, or participating in another clinical study.
4. Treatment with ultraviolet (UV) light (including tanning) during the previous 4 weeks.
5. Acute dermatitis outbreak on the arms or hands.
6. Subjects unable to comply with protocol restrictions
7. Subjects known to be unreliable or non-compliant with medical treatment, or unwilling to comply with multiple return visits.
8. Any condition or prior/present treatment, in the opinion of the investigators, should render the patient ineligible for the study
9. Known allergy to benzalkonium chloride or other ingredients in the fiteBac vehicle

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18-70 years of age, in generally good health with no significant underlying systemic disease requiring ongoing medications.
2. Hand eczema severity index (HECSI) with a score of greater than 50 (see Table 1 and reference 5)
3. Physician global assessment (PGA) of moderate to severe (with PGA severity scores graded as in Table 1 of reference 8: severe, moderate, mild, almost clear, clear).

Exclusion Criteria:

1. Topical corticosteroid or calcineurin inhibitor treatment during the last 7 days, prior to enrollment, on the hands and forearms
2. Systemic treatment with corticosteroids or other immunosuppressives during the last 14 days.
3. Subjects currently receiving (or received during the previous 4 weeks) other investigational drugs, treatments or devices, or participating in another clinical study.
4. Treatment with ultraviolet (UV) light (including tanning) during the previous 4 weeks.
5. Acute dermatitis outbreak on the arms or hands.
6. Subjects unable to comply with protocol restrictions
7. Subjects known to be unreliable or non-compliant with medical treatment, or unwilling to comply with multiple return visits.
8. Any condition or prior/present treatment, in the opinion of the investigators, should render the patient ineligible for the study
9. Known allergy to benzalkonium chloride or other ingredients in the fiteBac vehicle

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of fiteBac compared to emollient therapy | 1 month
  - To compare the efficacy of fiteBac skin care versus emollient therapy using standardized questionnaires, physical findings and photography over a one month treatment period in adults with hand dermatitis.

SECONDARY OUTCOMES:
Bacterial counts | 1 month
  - To compare the bacterial counts on the hands of patients with hand dermatitis treated with one month of fiteBac skin care versus emollient therapy
Physician Global Assessment | 1 month
  - To determine the Physician Global Assessment (PGA) of overall hand dermatitis severity with excellent response defined as clear or almost clear hands
Adverse events | 1 month
  - Number of adverse events on fiteBac versus emollient control
Number of flares | 1 month
  - To determine the number of flares on fiteBac versus emollient control
Number of study discontinuations | 1 month
  - To determine the number of study discontinuations on fiteBac versus emollient control
Patients Global Assessment score | 1 month
  - To determine the Patient's Global Assessment score on fiteBac versus emollient control

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States